CLINICAL TRIAL: NCT04539691
Title: Impacts of Static Magnetic Fields on Dysmenorrhea Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Southeastern University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2018-614-NSU
Record Dates: First submitted 2020-08-31; First posted 2020-09-07 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Period Pain
MeSH Terms: conditions — Dysmenorrhea

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Magnet and sham devices used weigh and look the same
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Magnet group (Experimental): Women wearing magnet
  a magnet, or sham device indistinguishable from the magnet (determined randomly), will be placed on her abdomen. If the pain is predominately in her abdomen, the device will be placed on the location with the most pain. If the pain is predominantly in the subjects back, the device will be placed on the lower abdomen on the midline between the umbilicus and the pubic bone.
  Interventions: Device: Magnet
- Sham group (Sham Comparator): Women wearing sham
  a magnet, or sham device indistinguishable from the magnet (determined randomly), will be placed on her abdomen. If the pain is predominately in her abdomen, the device will be placed on the location with the most pain. If the pain is predominantly in the subjects back, the device will be placed on the lower abdomen on the midline between the umbilicus and the pubic bone.
  Interventions: Device: Magnet

INTERVENTIONS:
Device: Magnet — Magnet or Sham is worn by subject in close proximity to their described maximum pain site

SUMMARY:
Study to determine the effectiveness of a certain type of magnet to reduce period pain

DETAILED DESCRIPTION:
Young women with their period pain levels of 6 or greater on a pain scale of 0-10 will wear a concentric magnet or a sham that is positioned close to the maximum pain site. The pain score after wearing either the magnet or sham will be recorded.

ELIGIBILITY:
Inclusion Criteria: Female with period pain score consistently equal to or greater than 6 on a pain scale of 0-10 -

Exclusion Criteria:

1. Pain not experienced on almost all menstrual cycles
2. Having secondary dysmenorrhea including endometriosis, fibroids or pelvic inflammatory disease
3. Having a pacemaker or any implanted wires or devices -

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Ages 18-35 years of age with period pain score consistently equal to or greater than 6 on a pain scale of 0-10
Enrollment: 60 (Actual)
Dates: Start 2018-08-30 (Actual); Primary Completion 2021-03-08 (Actual); Study Completion 2021-03-08 (Actual)

PRIMARY OUTCOMES:
Pain score scale of 1-10 / 1 being less pain 10 being more pain | 40 minutes
  Subject reported pain after wearing device

CONTACTS AND LOCATIONS:
Overall Officials: Harvey Mayrovitz, PhD, Principal Investigator — Nova Southeastern University
Locations (1):
- Nova Southeastern University, Davie, Florida, United States

IPD SHARING:
Plan to Share IPD: No